CLINICAL TRIAL: NCT02161926
Title: Dietary Restrictions Implications on Metabolic Changes in Obese Men : Comparison Between Two Groups of Different Ages (60-70 Years Old Versus 30-40 Years Old)
Brief Title: Assessments of Dietary Restrictions in Young and Elderly Obese Men : Metabolism Obesity Nutrition Age
Acronym: MONA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 13 149 03; 2013-A01543-42 (Other: RCB number)
Record Dates: First submitted 2014-06-06; First posted 2014-06-12 (Estimated); Last update posted 2018-01-05 (Actual); Status verified 2018-01

CONDITIONS: Obesity
Keywords: Obesity; dietary restrictions; metabolism; nutrition; elderly
MeSH Terms: conditions — Obesity | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- obese men from 60 to 70 years old (Experimental): Dietary restrictions in obese men (30<Body Mass Index<40 kg/m2)
  Interventions: Other: dietary restrictions
- obese men from 30 to 40 years old (Active Comparator): Dietary restrictions in obese men (30<Body Mass Index<40 kg/m2)
  Interventions: Other: dietary restrictions

INTERVENTIONS:
Other: dietary restrictions — Dietary restrictions during 8 weeks
  Other Names: Dietary restrictions (20 % dietary restrictions)

SUMMARY:
The prevalence of obesity is growing in elderly with heavy consequences in term of medical complications and mortality, so that this is nowadays an important public health issue.

The major therapeutic solution is dietary restrictions, but and the advantages and the metabolic consequences are not well known in elderly. The MONA study main aim is to assess the metabolic changes in this population, after dietary restrictions, compared to young people.

DETAILED DESCRIPTION:
Primary endpoint : Study the metabolic adaptations of the subcutaneous adipose tissue after a diet in elderly obese men compared to young obese men.

Secondary endpoints : Study the metabolic adaptations of skeletal muscle, the genetic adaptations of subcutaneous adipose tissue and skeletal muscle, the inflammatory and fibrosis modifications of subcutaneous adipose tissue, the insulinosensibility modifications, the modifications on the physical composition, modifications of the energy expenditure in resting state and the oxidation of the substrata, study the lipoproteins metabolism and identify new biomarkers. All those endpoints are studied comparing elderly obese subjects versus young obese subjects.

ELIGIBILITY:
Inclusion Criteria:

* 30 < years old < 40 OR 60 < years old < 70
* obesity : 30 < BMI < 40
* stable blood pressure (diastolic <90mmHg, systolic < 140mmHg)
* glycemia < 1,26g/L, LDL cholest <1,9-1,6g/L, Triglycerides <2,5g/L
* risk factors concerning high blood pressure, diabetes and dyslipidemia under control

Exclusion Criteria:

* Insulin dependent diabetes, non-insulin dependent diabetes
* high blood pressure
* dyslipidemia
* history of cardiovascular diseases or bariatric surgery
* undernutrition
* HbA1C >7%
* non authorized treatments : Glucagon-like peptide-1 agonists,
* incapacity to do physical activity

Ages: 30 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2014-05; Primary Completion 2016-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Lipolysis at resting and during physical activity test | Change after 8 weeks dietary restrictions
  Determine lipolysis at resting and during physical activity test by microdialysis, before dietary restrictions and after dietary restrictions (20% dietary restrictions)

SECONDARY OUTCOMES:
Metabolic parameters in skeletal muscle | Change after 8 weeks dietary restrictions
  To assess metabolic parameters before dietary restrictions and after dietary restrictions (20 % dietary restrictions)
Genetic markers | Change after 8 weeks dietary restrictions
  To assess genetic markers in adipose tissue and skeletal tissue before dietary restrictions and after dietary restrictions
Fibrosis and inflammatory markers in adipose tissue | Change after 8 weeks dietary restrictions
  To assess markers in adipose tissue before dietary restrictions and after dietary restrictions (20 % dietary restrictions)
insulinosensibility | Change after 8 weeks dietary restrictions
  To determine insulinosensibility before dietary restrictions and after dietary restrictions (20 % dietary restrictions)
Fat and muscles rates in the whole body | Change after 8 weeks dietary restrictions
  To determine fat and muscles rates by Dexa before dietary restrictions and after dietary restrictions
Energetic consumption | Change after 8 weeks dietary restrictions
  energetic consumption at resting and during physical activity, before dietary restrictions and after dietary restrictions
Lipoproteins metabolism | Change after 8 weeks dietary restrictions
  Before dietary restrictions and after dietary restrictions
biomarkers identification | Change after 8 weeks dietary restrictions
  New urinary and intestinal biomarkers identification, before dietary restrictions and after dietary restrictions

CONTACTS AND LOCATIONS:
Overall Officials: Claire Thalamas, MD PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France